CLINICAL TRIAL: NCT03725163
Title: Telepsychotherapy for the Treatment of Adolescents With Trichotillomania
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Michael Twohig, Ph.D., Professor, Utah State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9153
Record Dates: First submitted 2018-10-15; First posted 2018-10-30 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Trichotillomania
Keywords: Trichotillomania; Adolescents; Telepsychotherapy; AEBT; ACT
MeSH Terms: conditions — Trichotillomania

STUDY DESIGN:
Intervention Model Description: Participants will be randomized using block randomization to be assigned to a waitlist control condition or the treatment condition. Participants assigned to the waitlist control will have a 12-week waiting period prior to starting treatment. Those assigned to the treatment condition will begin therapy immediately.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): This arm will begin treatment immediately after completing the initial intake assessment.
  Interventions: Behavioral: Acceptance and Commitment Therapy Enhanced Behavior Therapy (AEBT)
- Waitlist Control (Other): Participants assigned to the waitlist control condition will begin a 12-week waiting period after completing the initial intake assessment before starting treatment.
  Interventions: Behavioral: Acceptance and Commitment Therapy Enhanced Behavior Therapy (AEBT)

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy Enhanced Behavior Therapy (AEBT) — This treatment approach blends traditional behavior therapy elements of habit reversal training and stimulus control techniques with the more contemporary behavioral elements of Acceptance and Commitment Therapy (ACT). The first phase of the treatment, clients are taught skills for stopping and preventing their unconscious pulling episodes. The second phase, clients are introduced to ACT. Unlike interventions that aim to change the type or frequency of pulling-related cognitions, this treatment uses strategies to change the function of these cognitions. Clients are taught to see urges for what they really are and to accept their pulling-related thoughts, feelings, and urges without fighting against them. Over the course of 10 session clients will learn to be aware of their pulling and warning signals, use self-management strategies for stopping and preventing pulling, stop fighting against their pulling-related urges and thoughts, and work toward increasing their quality of life.

SUMMARY:
The primary purpose of the current study is to evaluate the effectiveness of providing treatment for adolescents with trichotillomania through the use of telehealth. Parent or legal guardians' psychological flexibility scores will be assessed to determine if their levels of flexibility potentially moderate treatment outcomes.

The study will test the following hypotheses:

Hypothesis 1: Telepsychotherapy will result in significantly better trichotillomania symptom outcomes for adolescents than a waitlist control condition.

Hypothesis 2: Telepsychotherapy will result in significantly better psychological flexibility outcomes for adolescents than a waitlist control condition.

Hypothesis 3: Telepsychotherapy will result in significantly better overall wellbeing outcomes for adolescents than a waitlist control condition.

Hypothesis 4: Within-group changes (that include both conditions following treatment) will be significant from pre-treatment to post-treatment and will not significantly differ from post-treatment at 3, 6, and 12-month follow-up.

DETAILED DESCRIPTION:
The investigators of this study plan to recruit 60 participants, 30 adolescents and 30 parents or legal guardians. This number will provide adequate power (0.70) to detect a large effect size (d=.81). All portions of this study will be completed online using teleconferencing software, Zoom (similar to Skype).

Participants will be randomized into either a treatment or waitlist control group. All participants will receive treatment, however, those in the waitlist group will wait 12 weeks before beginning treatment. Treatment will consist of 10, 50 minute sessions with up to six short (10-15 minute) booster sessions during a three-month period following treatment. Participants and parents/guardians will complete full assessment batteries at intake, post-waitlist (only those in the waitlist condition), post-treatment, and 3, 6, and 12 months following treatment. Moreover, adolescent participants will be asked to track their daily pulling behavior each day while in treatment(with parent/guardian help if desired). This will be done through the use of daily text message reminders using app.eztexting.com to the parent/guardian that will include a link to the short (less then 5 minute) Qualtrics survey. All treatment sessions will take place online using video conferencing software (i.e., Zoom).

Parents/guardians will be invited to participate in the final 10 minutes of each session. This will allow for the adolescent to review what they have learned and also allow the parent/guardian to be involved in the fulfillment of treatment goals and to assist with skill-building throughout the week. Parents will also be give a short (1/2 to 1 page) handout following each session that will explain what was taught and how they can best help the participant make progress. Parents will also be asked to complete a short measure of psychological flexibility at intake, post-waitlist (only when applicable), post-treatment, and 3, 6, and 12-months following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meet DSM-5 criteria for trichotillomania.
* Seeking treatment primarily for trichotillomania-related concerns.
* 12-17 years old.
* Reside in Utah.
* Speak fluent English.

Parents:

* Must be fluent English speaker.

Exclusion Criteria:

* Currently receiving psychotherapy.
* Started or changed psychotropic medication in the past 30 days.
* Planning to start or change psychotropic medication during the course of the current study.
* Completed high school.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2020-08-05 (Estimated); Study Completion 2020-08-05 (Estimated)

PRIMARY OUTCOMES:
Trichotillomania Scale for Children-Chile and Parent Versions (TSC-C & TSC-p) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  This self-report measure can be filled out by both the adolescent and parent. This measure is broke into 2 components: severity (5 items) and distress/impairment (7 items). A total of 3 scores are obtained, one for each component and a total score. This measure provides information about symptom severity and level of impairment or distress of trichotillomania for the client. Items 1-5 represent the severity score, each item is scored 0-2 with 2 representing higher severity. Items 1-5 are summed then divided by 5 to give a severity score. Items 6-12 represent the Distress/Impairment section and follow a similar scoring format summing each item and dividing by 7 to represent the Distress/Impairment score. The Severity Score and Distress/Impairment score are summed to give a total score. The minimum value for scores can be 0, with the highest score being 4 for the total score.
Acceptance and Action Questionnaire for Trichotillomania (AAQ-TTM) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  This measure assesses a participant's overall levels of psychological inflexibility in relation to trichotillomania and how impairing trichotillomania may be for the individual. Each item ranges on scores from 1 (Never true) to 7 (always true). Higher scores on each item indicate higher levels of distress or psychologically inflexibility in relation to their trichotillomania. The values for each items are summed to provide a total score. Higher scores tend to indicate greater psychological flexibility. Items 2,3,4,5,7,8, and 9 are reversed scored.
Warwick-Edinburgh Mental Well-being Scale (WEBWMS) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  This is a 14-item Likert-type scale that measures overall well-being for participants. Each item has scores ranging from 1="None of the time" to 5 "All of the time". Higher scores indicate higher levels of overall well-being for a client.

SECONDARY OUTCOMES:
Acceptance and Fusion Questionnaire for Youth (AFQ-Y8) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  The AFQ-Y measures psychological acceptance, cognitive fusion, and similar processes related to Acceptance and Commitment Therapy model. It serves as a potential predictor of negative outcomes.This is an 8-item Likert-type scale, with values ranging from 0= "Not at all True" to 4= "Very True". Scores from each item are summed and divided by the total number of items completed, then this average score is multiplied by 8. Higher scores indicate greater levels of distress or impairment.
Youth Outcome Questionnaire (YOQ-C & YOQ-P) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  The YOQ covers a variety of situations, moods, and behaviors which are common to adolescents and these may or may not apply to each participant. It provides an assessment for tracking adolescent behavior by both the adolescent and parent and gives an understanding of the effectiveness of therapy. This is a 35-item Likert-type scale with items 1-30 ranging from 0 = "Never or Almost Never" to 4 = "Always or almost always", while items 31-35 range from 0 = "Haven't met therapist yet" to 5 = "Strongly agree". The first 30 items indicate total distress in a clients' life. Scores greater than or equal to 46 indicate clinically significant distress or impairment.
Parental Acceptance Questionnaire (6-PAQ) | Changes in scores from baseline, 10-week post-treatment, and 3-, 6-, and 12-month follow-ups will be assessed.
  The 6-PAQ provides a measure of psychological flexibility for parents/legal guardians in their interactions with their children and parenting behaviors. This is an 18-item Likert-type scale with responses ranging from 1 = "Strongly disagree/never" to 4 = "Strongly agree/almost always". Items 1, 2, 5, 7, 10, 15, and 18 are reverse scored. Lower scores represent greater levels of parental psychological flexibility, while higher scores indicate greater levels of parental psychological inflexibility.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Twohig, PhD, Principal Investigator — Utah State University
Locations (1):
- Utah State University, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided
Once the study is complete it is possible that we may share deidentified data from participant survey scores, the protocol used, and the consent form used for the study.